CLINICAL TRIAL: NCT01214291
Title: Phase III Randomized, Double-Blind, Placebo Controlled, Multicenter Efficacy and Safety Study of Toremifene Citrate 80 mg for the Reduction in the Risk of New Bone Fracture Occurrences in Men With Prostate Cancer on Androgen Deprivation Therapy
Brief Title: Efficacy and Safety Study of Toremifene Citrate for the Reduction in the Risk of New Bone Fracture Occurrences in Men With Prostate Cancer
Acronym: TREAT2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: cost of conducting the study and increased burden on the clinical trial professionals make it impossible for us to proceed with the development of the drug.
Sponsor: GTx (Industry)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: G300213
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Risk of Bone Fracture Occurrences
Keywords: fractures; prostate cancer; androgen deprivation therapy
MeSH Terms: conditions — Fractures, Bone; Prostatic Neoplasms | interventions — Toremifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Toremifene — Toremifene 80mg daily

SUMMARY:
The purpose of this study is to determine whether Toremifene Citrate is effective in reducing the risk of bone fractures in men with prostate cancer who are on Androgen Deprivation Therapy.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary signed informed consent
* have histologically documented prostate cancer
* have been on ADT treatment for 6 months prior to randomization or intermittent LHRHa for preceeding 12 months
* expected to continue LHRHa therapy uninterrupted for the next 12 months
* have total testosterone levels less than 50 ng/dL
* Have BMD of lumbar spine or femoral neck at or below the BMD thresholds
* have a Zubrod performance status <or equal to 1
* subject weight <300 lbs(<136 kg)
* agree to complete a daily diary of medication intake
* agree not to take excluded medications throughout the trial
* agree to use an effective method of contraception
* have adequate bone marrow, liver and renal functions

Exclusion Criteria:

* Currently or previously exposed
* within the past 5 years to intravenous bisphosphonates, strontium ranelate or Denosumab
* for more than 3 years to oral bisphosphonates
* within the last 45 days to PTH or PTH derivative, anabolic steroids or testosterone, SERMs, calcitonin, calcitriol or oral gluccorticoids
* have any disease or condition that would preclude an accurate evaluation of radiographs of the thoracic or lumbar spine
* have <8 evaluable vertebrae
* have a BMD T score <-4 at the lumbar spine or total hip or femoral neck
* have any history of other carcinomas within the last 5 years
* Serum PSA > 5ng/mL at baseline under ADT
* have Paget's disease, Cushing's disease, chronic hepatitis or cirrhosis or rheumatoid arthritis
* have active uncontrolled systemic viral, bacterial or fungal infections
* have a clinically significant concurrent illness or psychological, familial, sociological, geograhical or other condition that would not permit adequate follow-up and compliance
* received treatment with other investigational agents within 30 days
* taking finasteride, dutasteride, danazol or testosterone like substances
* taking herbal medicines or dietary supplements
* have a history of thromboembolic disease including DVT or pulmonary embolus
* have a QTcF of > or equal to 450 msec or congenital or acquired QTc prolongation
* have HIV
* calcicum urolithiasis prohibiting the use of vitamin D

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To confirm the efficacy of toremifene 80mg compared with placebo in the reduction in the risk of new bone fracture occurrences in men with prostate cancer on androgen deprivation therapy as measured by semiquantitative assessment of vertebral fractures | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Steiner, MD, Study Director — GTx
Locations (1):
- VA Puget Sound, Seattle, Washington, United States